CLINICAL TRIAL: NCT04468412
Title: Influence of COVID-19 on Vascular Endothelial Function
Acronym: COVAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Bernhoven Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL2020-6555
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-09

CONDITIONS: COVID; Vascular; Damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Carotid Artery Reactivity Testing — The carotid artery reactivity (CAR) test assesses macrovascular endothelial function by measuring the carotid artery diameter in response to sympathetic stimulation. Participants are in the supine position with the neck extended for assessment of the carotid artery. Left carotid artery diameter is recorded continuously during baseline (30 seconds) and during immersion of the right hand up to the wrist in icy water (4°C) for 3 minutes. CAR can either represent a dilatory response (normal endothelial function) or a constrictive response (endothelial dysfunction) of the carotid artery.
  Other Names: Cold pressor test

SUMMARY:
Rationale: Infection with severe acute respiratory syndrome coronavirus (SARS-CoV) 2 could result in endothelial dysfunction with increased risk of arterial thrombotic events by downregulating the expression of angiotensin converting enzyme 2 (ACE2). Endothelial function can be easily and non-invasively determined by carotid artery reactivity (CAR) testing.

Objective: To investigate the predictive value of endothelial dysfunction, measured by carotid artery reactivity testing, for 1-year cardiovascular events in patients with past COVID-19 infection.

Study design: A prospective observational longitudinal cohort study.

Study population: Patients recovered from confirmed infection with SARS-CoV2.

Main study parameters/endpoints: macrovascular endothelial function measured by carotid artery reactivity testing.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV2 infection by polymerase chain reaction on nasopharyngeal swab, sputum or bronchoalveolar lavage.
* At least 6 and no more than 20 weeks after resolution of COVID-19 related symptoms
* ≥ 16 years old

Exclusion Criteria:

* Recent (<3 months) angina pectoris, myocardial infarction, stroke, or heart failure
* Raynaud syndrome, scleroderma, complex regional pain syndrome of the upper extremity or presence of arteriovenous fistula or open wounds on both the upper extremities.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with past COVID-19 infection will be recruited at Bernhoven hospital, the Netherlands.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial dysfunction | CAR will be measures between 6 and 20 weeks and 1 year after recovery from COVID-19.
  Change in endothelial dysfunction as determined by CAR test.

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 year
  MACE include non-fatal myocardial infarction, non-fatal ischemic stroke, acute limb ischemia, need for revascularization, amputation and cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel C Warle, PhD, Principal Investigator — Radboud University Medical Center; Andre S van Petersen, PhD, Principal Investigator — Benhoven
Locations (1):
- Bernhoven, Uden, Netherlands

IPD SHARING:
Plan to Share IPD: No